CLINICAL TRIAL: NCT06798727
Title: Evaluation Safety and Explore Efficacy Long-term Follow-up Study on Subjects Receiving SMUP-IA-01 or Active Control
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-SMUP-IA-01-P02-F/U
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
Keywords: human umbilical cord blood derived mesenchymal stem cells; hUC-MSCs; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Phase 2's long term follow-up Study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMUP-IA-01(low-dose) (Experimental): A single knee administration of SMUP-IA-01 (low-dose, 4.0 x 10^6 cells/2mL) (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(low-dose)
- SMUP-IA-01(mid-dose) (Experimental): A single knee administration of SMUP-IA-01 (mid-dose, 1.0 x 10^7 cells/2mL) (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(mid-dose)
- High Hyal Plus Inj. (Active Comparator): A single knee administration of High Hyal Plus Inj.(1% Sodium Hyaluronate 20mg/2ml)
  Interventions: Drug: High Hyal Plus

INTERVENTIONS:
Biological: SMUP-IA-01(low-dose) — A single knee administration of SMUP-IA-01(low-dose, 4.0 x 10^6 cells/2mL)
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: SMUP-IA-01(low-dose)
Biological: SMUP-IA-01(mid-dose) — A single knee administration of SMUP-IA-01(mid-dose, 1.0 x 10^7 cells/2mL)
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: SMUP-IA-01(mid-dose)
Drug: High Hyal Plus — A single knee administration of Hyaluronic acid(1% Sodium Hyaluronate 20mg/2ml)
  Arms: High Hyal Plus Inj.

SUMMARY:
This is a follow-up study to investigate the long-term safety and explore efficacy of SMUP-IA-01, for the treatment of Knee Osteoarthritis. Subjects who participated in and completed the initial stage of the Phase II trial (NCT05182034) will be followed-up until 60 months.

DETAILED DESCRIPTION:
The subjects will be followed up at 12-month, 24-month, 36-month, 48-month and 60-month after the initial administration of SMUP-IA-01.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who completed the safety and explore efficacy evaluations in SMUP-IA-01 Phase II clinical trial.
2. Subject who voluntarily decided to participate and signed the consent form after receiving explanations on the clinical trial.

Exclusion Criteria:

1. Subject who were not enrolled in phase II clinical trial of SMUP-IA-01 for assessing safety and explore efficacy.
2. Other subjects, excluding those listed above, who were deemed unsuitable by the PI

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of total score in WOMAC (Western Ontario and McMaster University) | Time Frame: Month 12, 24, 36, 48 and 60 after treatment
  Comparing WOMAC total score changes with baseline scores of SMUP-IA-01 phase I trial and scores of f/u study at 12 months, 24 months, 36 months, 48 months and 60months after treatment (score range 0-96, higher score represent worse symptoms).

SECONDARY OUTCOMES:
Change of score in WOMAC three subscales (Pain, stiffness, physical function) aginst MP-SMUP-IA-01-P02's baseline. | Time Frame: Month 12, 24, 36, 48 and 60 after treatment
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
Change of score in 100 mm VAS (Visual Analogue Scale) | Time Frame: Month 12, 24, 36, 48 and 60 after treatment
  The score ranges from "0" or no pain to "100" very severe pain
Change of score in IKDC(International Knee Documentation Committee) | Time Frame: Month 12, 24, 36, 48 and 60 after treatment
  The scores for each category are summed up and divided into 87, which is the maximum score possible, and then is evaluated by converting it into a scale of 100 points. Higher score indicates better function and less symptoms for the knee.
Change of score in WORMS(Whole-Organ Magnetic Resonance iMaging Score) | Time Frame: Month 12 and 24 after treatment
  For structural and tissue evaluation of knee, MRI image of detailed knee parts are graded from min. 0 to max. 6. Lower number indicate normal status
Change in K&L(Kellgren-Lawrence) grade | Time Frame: Month 12, 24 and 60 after treatment
  The K & L grade is 0 to 4 Grade, which means that the higher the grade, the greater the joint damage and the stenosis of the joint
Change in joint space width | Time Frame: Month 12, 24 and 60 after treatment
  Evaluation of disease progression in target knee as ascertained by change from baseline in joint space width (JSW) determined using radiography
Change in mechanical axis, anatomical axis | Time Frame: Month 12, 24 and 60 after treatment
  The degree of deformation of the lower half of the body is measured by measuring the angles of the mechanical axis and the anatomical axis with respect to the vertical axis. Mechanical axis: A line connecting the femoral head center point and the ankle joint center point. Anatomical axis: The middiaphyseal line of the femur and tibia

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Seoul Nation University Bundang Hospital, Gyeonggi-do
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospita, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No